CLINICAL TRIAL: NCT04665011
Title: Validation of Indicor Photoplethysmography (PPG) Valsalva Pulse Response vs Non-invasive Blood Pressure
Status: Completed | Type: Observational
Sponsor: Vixiar Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: PROT 000054
Record Dates: First submitted 2020-12-08; First posted 2020-12-11 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Clinically stable adults, including heart failure patients visiting an outpatient clinic: Observational to compare simultaneous pulse tracings from PPG and non-invasive blood pressure monitors in capturing the pulse responses to a Valsalva maneuver.
  Interventions: Device: Indicor; Device: Caretaker

INTERVENTIONS:
Device: Indicor — A simple, non-invasive tool to report pulse response to a Valsalva maneuver
Device: Caretaker — non-invasive blood pressure monitor

SUMMARY:
This study designed is compare the pulse response to the Valsalva maneuver between a photoplethysmography sensor (PPG) and non-invasive blood pressure sensor for the purpose of validating the PPG methodology in deriving a value for the Valsalva pulse response. The aim is to show that the PPG method captures the same phase responses as the blood pressure monitor and the primary outcome is the correlation between pulse amplitude ratios for the pulse at the end of the Valsalva to an average baseline pulse.

DETAILED DESCRIPTION:
With both a photoplethysmography (PPG; Indicor, Vixiar Medical,. Baltimore, MD) and non-invasive blood pressure (Caretaker, Caretaker Medical, Charlottesville, VA) sensors in place on the index and middle fingers, respectively, each patient will be asked to perform three mild, 10-sec Valsalva maneuvers with at least 45 seconds between. Pulse recordings will be collected from each device to compare phases of the Valsalva pulse response including pulse amplitude changes and baseline movement. The primary outcome is the correlation between pulse amplitude ratios for the pulse at the end of the Valsalva to an average baseline pulse.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable adults, including heart failure patients visiting an outpatient clinic

Exclusion Criteria:

* Atrial flutter or atrial fibrillation with an irregular ventricular response
* Significant atrial or ventricular ectopy
* History of paradoxical emboli
* Hypertrophic obstructive cardiomyopathy
* Known intracardiac shunt
* Known severe aortic valve stenosis
* Known severe mitral valve stenosis
* History of embolic CVA
* Myocardial infarction within one week of intended Indicor testing
* Uncontrolled hypertension (systolic BP >160mmHg or diastolic BP>100mmHg)
* Hypotension (systolic BP <90mmHg)
* Symptomatic bradycardia
* Known cholesterol emboli
* Poor left ventricular function with left ventricular thrombus
* Unstable angina
* Significant aortic valvular disease
* Patients weighing less than 40kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study sample has a focus on heart failure patients as this is a clinical target population for the clinical use of the Indicor. However, non-heart failure subjects may be needed to ensure that a range of normal outcome values are included in the analysis. Therefore, at least 70% of the enrollment is intended to be derived from a cardiology practice office, and up to 30% of the enrollment may be non-patient participants.
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-01-28 (Actual); Study Completion 2021-01-28 (Actual)

PRIMARY OUTCOMES:
pulse amplitude ratio | 5 minutes
  The correlation between PPG-based and non-invasive blood pressure pulse amplitude ratio during a Valsalva maneuver.

SECONDARY OUTCOMES:
Phases of valsalva pulse response | 5 minuntes
  The agreement between PPG-based and non-invasive blood pressure pulse tracings during a Valsalva maneuver.

CONTACTS AND LOCATIONS:
Overall Officials: Keith H. Newby, M.D., Principal Investigator — Fort Norfolk Cardiology Associates
Locations (1):
- Fort Norfolk Cardiology Associates, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No